CLINICAL TRIAL: NCT04368143
Title: COVID-19 Immune Repertoire Sequencing
Acronym: IMSEQ
Status: Completed | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Other Study IDs: IMSEQ
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: COVID; SARS-CoV 2; Corona Virus Infection; RDT; B Cell
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This concerns a single-center prospective interventional cohort study. Laboratory-confirmed COVID-19 patients will be asked to donate blood at at least two different timepoints. This will allow us to investigate T and B cell evolutions during the course of infection and recovery. The expected duration of the study is four months or the total duration of the SARS-CoV-2 circulation in Belgium (whichever is shortest).

ELIGIBILITY:
Inclusion Criteria:

* laboratory confirmed COVID-19 acute infection
* be older than 18 years of age
* be hospitalized at the UZA
* willing and able to provide written informed consent by the participant or its legal representative (for instance in case of medical incapacitation)

Exclusion Criteria:

* younger than 18 years old
* Ambulatory patients

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in an in-patient hospital setting. Patients will be recruited at UZA, where SARS-CoV-2 infected individuals might present. Patients with (mild) respiratory complaints and suspected risk of having contracted SARS-CoV-2 (risk contact with confirmed case, travel history to endemic area) will be tested and isolated in awaiting laboratory SARS-CoV-2 test results. In case of mild respiratory complaints, people will be discharged immediately for home isolation; while patients in need for hospital care will be hospital-admitted (in isolation rooms). If SARS-CoV-2 test results return positive, these hospitalized patients will be asked to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
provide proof-of-concept that (longitudinal) B cell repertoire mining allows identification of emerging virus specific B cell receptor variable regions. | 4 months

SECONDARY OUTCOMES:
study evolutions in B and T cell repertoires to understand COVID-19 specific immune responses fundamentally. | every 7 days during hospitalization a bloodsample is taken
clinical and epidemiological description of UZA hospitalized COVID-19 patients | at hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Universitairy hospital of Antwerp, Antwerp, Belgium